CLINICAL TRIAL: NCT01681043
Title: Sleep Investigation in Respirator Treated ICU Patients: the Importance of Intensive Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Principal Investigator, Yuliya Boyko, MD, Vejle Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: S-20120001
Record Dates: First submitted 2012-08-23; First posted 2012-09-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Sleep
Keywords: Sleep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24 hour PSG under ordinary conditions (No Intervention): 24 hour PSG in 46 patients under ordinary (routine) conditions
- 24 hours PSG under protocol 'Quiet in the room' (Active Comparator): 24 hour PSG in the same 46 patients with protocol 'Quiet in the room' from 10 p.m. til 6 a.m.
  Interventions: Behavioral: protocol 'Quiet in the room'

INTERVENTIONS:
Behavioral: protocol 'Quiet in the room' — Protocol 'Quite in the room' between 10 p.m. and 6 a.m.
  * nurse nearby
  * no visits after 10 p.m.
  * decreased alarm sound in ventilator and monitor
  * decreased light intensity
  * no unnecessary conversations around the patient
  * medication should be limited to max 1-2 times in this time period
  * no unnecessary therapeutic or diagnostic procedures in this time period
  * earplugs and sleep masks
  Arms: 24 hours PSG under protocol 'Quiet in the room'

SUMMARY:
Sleep investigation in respirator treated ICU patients: the importance of intensive environment.

Sleep disturbances in the ICU seem to lead to development of delirium, prolonged ICU stay and increased mortality.

The hypothesis of this study is: minimizing of disturbing factors in the ICU, such as noise, light, therapeutic and diagnostic procedures between 10 p.m. and 6 a.m. will improve sleep quality in respirator treated ICU patients.

Methods: randomized interventional study. 48-hour polysomnographic sleep measurement acc. AASM's standard in 46 awake respirator treated patients: 24 hours under ordinary circumstances and 24 hours under the protocol 'Quiet in the room' between 10 p.m. and 6 a.m. after randomization.

ELIGIBILITY:
Inclusion Criteria:

* awake and relevant respirator treated patients with expected 2 or more respirator dags

Exclusion Criteria:

* GCS < 11
* cerebral hemorrhage or infarction during the current hospitalization
* delirium
* inotropes and/or vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
the number of arousals | per hour of sleep
  arousals will be scored during the sleep periods and the index - arousals per hour of sleep - will be counted

SECONDARY OUTCOMES:
total sleep time | 24 hours
  total sleep time during 24 hour period
N1 sleep | 24 hours
  N1 sleep stage will be scored during sleep periods (dag sleep/night sleep)and the percent of N1 sleep will be counted
N2 sleep | 24 hours
  N2 sleep stage will be scored during sleep periods and the percent of N2 sleep will be counted
N3 sleep | 24 hours
  N3 sleep stage will be scored during sleep periods and the percent of N3 sleep will be counted
REM sleep | 24 hours
  REM sleep will be scored during sleep periods and the percent of REM sleep will be counted

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia and Intensive Care, Vejle Hospital, Vejle, Denmark